CLINICAL TRIAL: NCT06169605
Title: Assessment of the Effect of Tumor Thickness and Site on Level IV Cervical Lymph Nodes in Squamous Cell Carcinoma of the Tongue and Floor of the Mouth: A Case Series Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Shawky, Assistant lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cairo uni PhD
Record Dates: First submitted 2023-12-03; First posted 2023-12-13 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Tongue Neoplasms
MeSH Terms: conditions — Tongue Neoplasms | interventions — Neck Dissection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with squamous cell carcinoma of the tongue and floor of the mouth (Experimental): Intervention group
  Interventions: Procedure: removal of primary tumor, neck dissection

INTERVENTIONS:
Procedure: removal of primary tumor, neck dissection — removal of the primary tumor with safety margins and removal of the neck lymph node levels I, II, III and IV. histological assessment of tumor thickness and whether it is associated with positive nodes in level IV or not.

SUMMARY:
Regarding oral cavity cancer, the high incidence of neck metastasis along with its impact on survival and prognosis are in favor of elective neck dissection. Moreover, occult metastases could develop at lower levels in the neck (levels IV-V) Regarding the tongue, the rate of skip (occult) metastasis involving unremoved level IV cervical lymph nodes in squamous cell carcinoma of the tongue ranges from 0 % - 11.4 %. However, no data is available or a correlation between the risk of level IV involvement and the affection of specific tongue subsites or a certain cutoff value of tumor thickness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with squamous cell carcinoma of the tongue and floor of the mouth.
* Age group: from 15 to 60 years old
* No sex predilection

Exclusion Criteria:

* Patients with recurrent squamous cell carcinoma of the tongue and floor of the mouth.
* Irradiated patients or those taking chemotherapy.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
tumor thickness in mellimeters | one week: specimens are submitted immediately after surgery
  histological assessment of tumor thickness of the resected tumor and assessment of level IV lymph nodes
Number of affected level IV cervical lymph nodes | One week : submitted immediately after surgery
  In each case the specimen will be assessed for level IV lymph nodes affection

SECONDARY OUTCOMES:
affected tongue site in relation to level IV cervical lymph nodes | One week
  histological assessment of level IV lymph nodes to determine if it is affected with tumor site on the tongue (lateral border, dorsum, ventral ....) which will be documented before surgery during examination

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shawky, MSc, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
will be available upon reasonable request
Supporting Information: Study Protocol, SAP
Time Frame: After study completion
Access Criteria: From Corresponding author

REFERENCES:
- [Background] Fakih AR, Rao RS, Borges AM, Patel AR. Elective versus therapeutic neck dissection in early carcinoma of the oral tongue. Am J Surg. 1989 Oct;158(4):309-13. doi: 10.1016/0002-9610(89)90122-0. PMID 2802032
- [Background] Kligerman J, Lima RA, Soares JR, Prado L, Dias FL, Freitas EQ, Olivatto LO. Supraomohyoid neck dissection in the treatment of T1/T2 squamous cell carcinoma of oral cavity. Am J Surg. 1994 Nov;168(5):391-4. doi: 10.1016/s0002-9610(05)80082-0. PMID 7977957
- [Background] Hutchison IL, Ridout F, Cheung SMY, Shah N, Hardee P, Surwald C, Thiruchelvam J, Cheng L, Mellor TK, Brennan PA, Baldwin AJ, Shaw RJ, Halfpenny W, Danford M, Whitley S, Smith G, Bailey MW, Woodwards B, Patel M, McManners J, Chan CH, Burns A, Praveen P, Camilleri AC, Avery C, Putnam G, Jones K, Webster K, Smith WP, Edge C, McVicar I, Grew N, Hislop S, Kalavrezos N, Martin IC, Hackshaw A. Nationwide randomised trial evaluating elective neck dissection for early stage oral cancer (SEND study) with meta-analysis and concurrent real-world cohort. Br J Cancer. 2019 Nov;121(10):827-836. doi: 10.1038/s41416-019-0587-2. Epub 2019 Oct 15. PMID 31611612
- [Background] Shah JP, Candela FC, Poddar AK. The patterns of cervical lymph node metastases from squamous carcinoma of the oral cavity. Cancer. 1990 Jul 1;66(1):109-13. doi: 10.1002/1097-0142(19900701)66:13.0.co;2-a. PMID 2354399
- [Background] Dias FL, Lima RA, Kligerman J, Farias TP, Soares JR, Manfro G, Sa GM. Relevance of skip metastases for squamous cell carcinoma of the oral tongue and the floor of the mouth. Otolaryngol Head Neck Surg. 2006 Mar;134(3):460-5. doi: 10.1016/j.otohns.2005.09.025. PMID 16500445
- [Background] Matos LL, Manfro G, Santos RV, Stabenow E, Mello ES, Alves VA, Pinto FR, Kulcsar MA, Brandao LG, Cernea CR. Tumor thickness as a predictive factor of lymph node metastasis and disease recurrence in T1N0 and T2N0 squamous cell carcinoma of the oral tongue. Oral Surg Oral Med Oral Pathol Oral Radiol. 2014 Aug;118(2):209-17. doi: 10.1016/j.oooo.2014.03.023. Epub 2014 Apr 12. PMID 24906946